CLINICAL TRIAL: NCT00473850
Title: Establishing the Genetic Profile of Multiple Hereditary Exostoses (HME) in Families of BC
Status: Terminated | Type: Observational
Why Stopped: This study is recruiting under a different title - "Genotype-Phenotype Correlation of Multiple Hereditary Exostoses: Multicentre Project" NCT00474331
Sponsor: University of British Columbia (Other)
Collaborators: Circle of Care (Unknown); Vancouver Foundation (Other); Children's & Women's Health Centre of British Columbia (Other)
Responsible Party: Dr. Christine Alvarez, University of British Columbia
Other Study IDs: H98-70441
Record Dates: First submitted 2007-05-14; First posted 2007-05-16 (Estimated); Last update posted 2011-04-15 (Estimated); Status verified 2011-04

CONDITIONS: Exostoses, Multiple Hereditary
Keywords: DNA sequencing; EXT genes; Hereditary Multiple Exostoses,; also known as Multiple Hereditary Exostoses,; also known as Hereditary Multiple Osteochondromas
MeSH Terms: conditions — Exostoses, Multiple Hereditary

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective

SUMMARY:
The purpose of this study is to establish the genetic profile of families in British Columbia with HME.

DETAILED DESCRIPTION:
The purpose of this study is to establish the genetic make-up of families and patients with HME. This will occur as the patient presents to a regular clinic visit. Dr. Alvarez will be introduced to interested patients and their parent(s) and a brief discussion about the project will occur. If the patient and their direct family are interested they will be entered into the study. This will involve interviewing the patients and their direct family. This interview will take about 1 hour. We are interested in identifying all affected family members as far up the family tree as possible. We ask that the idea of the study be introduced to extended family members by the participating family members and then have them call Dr. Alvarez to set up an appointment. Each available member will be interviewed and a physical exam done to determine the location of osteochondromas. In addition, Xrays will be done to determine the location of all osteochondromas. All Xrays will be reviewed. No new ones will be taken unless it is part of the patient's routine care.

To complete the genetic work up DNA analysis will be done on all available family members. This will entail obtaining a blood sample from each family member willing to partake in the study. These blood samples will be used only for the purpose of identifying abnormalities in the genes related to osteochondromas. The blood samples will be taken at British Columbia's Children's Hospital and processed there. DNA samples will be kept confidential.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with HME

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Benetic profile of families in British Columbia with HME.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 1998-12; Study Completion 2023-03 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Christine Alvarez, MD, Principal Investigator — University of British Columbia
Locations (1):
- BC Children's Hospital, Vancouver, British Columbia, Canada